CLINICAL TRIAL: NCT03146637
Title: Phase II Randomized Comparison Clinical Trial of Target Activated CIK for Advanced Liver Cancer
Brief Title: Study of Activated CIK Armed With Bispecific Antibody for Advanced Liver Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benhealth Biopharmaceutical (Shenzhen) Co., Ltd. (Industry)
Collaborators: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BK2016.01
Record Dates: First submitted 2017-05-02; First posted 2017-05-10 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Advanced Liver Cancer
Keywords: Activated CIK; MUC1/CEA/EpCAM/GPC3; Bispecfic antibody; liver cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a phase II clinical trial of single-center, randomized (1:1of targeted activation CIK and traditional CIK therapy ).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: With the method of minimum randomized dynamic random by the interactive network response system (IWRS),Participants were randomly assigned to two groups,receive activated CIK or activated CIK armed with anti-CD3-MUC1/CEA/EpCAM/GPC3 bispecific antibody,every participant has a unique identification number and emergency letter which have the information of group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activated CIK armed with bispecific antibody treatment group (Experimental): CIK cells were activated by bispecific antibody of anti-CD3-MUC1/CEA/EpCAM/GPC3
  Interventions: Biological: Activated CIK
- Traditional CIK treatment group (Active Comparator): CIK cells were not activated
  Interventions: Biological: CIK

INTERVENTIONS:
Biological: Activated CIK — Activated CIK armed with bispecific antibody were infused for 3 days，after 2 days，bispecific antibody was infused separately for 3 days
  Arms: Activated CIK armed with bispecific antibody treatment group
Biological: CIK — Traditional CIK were infused for 3 days
  Arms: Traditional CIK treatment group

SUMMARY:
This is a phase II Randomized comparison clinical trial of activated CIK armed with anti-CD3-MUC1/CEA/EpCAM/GPC3 bispecific antibody for advanced liver cancer. And the aim of this research is to study the clinical efficacy and safety of activated CIK armed with anti-CD3-MUC1/CEA/EpCAM/GPC3 bispecific antibody for liver cancer.

DETAILED DESCRIPTION:
Liver cancer is one of the most common malignancies in China, ranking fourth in all malignant tumors and third in mortality. Immunetherapy is considered to be one of the most promising means of human against cancer. This is a phase II clinical trial of single-center, randomized (1:1of targeted activation CIK and traditional CIK therapy )comparison clinical trial of activated CIK armed with anti-CD3-MUC1/CEA/EpCAM/GPC3 bispecific antibody for advanced liver cancer. The investigators plan to recruit for 80 cases patients with advanced liver cancer, the first 20 cases were directly received treatment of activated CIK, and the cases after the 20th were randomly assigned to two group，one of the two group will receive treatment of traditional CIK, and the other receive activated CIK. The result of this study was statistic and analysed with the record of Response Evaluation Criteria In Solid Tumors(RECIST1.1) evaluation standard.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old;
2. The patient is diagnosed as advanced liver cancer,MUC1/CEA/EpCAM/GPC3 is positive;
3. There is at least one tumor should be measured,and length≥10mm of focus not at lymph node or length≥10mm of focus at lymph node;
4. C interval of BCLC;
5. The patient can't tolerate system(systemic chemotherapy/molecular targeted therapy) or local therapies;
6. Child-Pugh Score ≤7;
7. If the patient received adjuvant chemotherapy after local treatment,the time should be more than 4 weeks after the end of chemotherapy, and disease progression or metastasis patients can also assigned into the group;
8. The time of surgical treatment≥ 3 months ;At the end of the intervention, radiotherapy and the end of the ablation time is more than 4 weeks;
9. The expected survival time ≥4 months；
10. The patient did not took any antitumor drugs within two weeks(any antitumor drugs, Chinese patent medicine including Delisheng injection, Kanglaite injection, Aidi injection, huaier granule and Ganfule Pian);
11. ECOG Score ≤1；
12. HBV DNA<10^4copies/ml（2000IU/ml);
13. Serum albumin≥28g/L,ALT and AST≤5.0×ULN,TBIL≤1.5×ULN, electrolyte is normal, proteinuria = 0 ~ 1 +, serum creatinine≤1.5 x ULN;
14. Tests of blood,liver and kidney should meet the following criteria:WBC≥3×10^9/L,NEUT≥1×10^9/L,Hemoglobin ≥90 g/L,ANC≥1.5×109/L,PLT≥50×10^9/L;
15. No serious disease are conflicts with the solution(such as autoimmune disease,immunodeficiency,orgen transplantation);
16. Sign the informed consent;

Exclusion Criteria:

1. Severe cirrhosis, medium or above ascites;
2. Cancer embolus in the main portal vein and first branch, Hepatic duct and first branch, hepatic vein, inferior vena cava;;
3. Patients of T cell lymphoma、myeloma,and patients are using immunosuppressant;
4. Systemic autoimmune diseases, allergic constitution or immunocompromised patients.
5. Patients of chronic diseases need immune stimulant or hormone therapy ;
6. Patients of active bleeding or coagulant function abnormality（PT>16s、APTT>43s、TT>21s、INR≥2）,and patients of bleeding tendency or are receiving thrombolysis and anticoagulation and antiplatelet therapy;
7. Women who is pregnant or during breast feeding or plan to pregnant in 2 years,and not willing to contraception during the test;
8. Any significant clinical and laboratory abnormalities, the researchers think that affect the safety, such as: incontrollable active infection (> NCI - CTC AE v4.0 standard level 2), uncontrolled diabetes (> level 2 of NCI - CTC AE v4.0 ), hypertension and can't be controlled by two or less hypotensor(systolic pressure < 140 mmHg, diastolic pressure < 90 mmHg), grade II or above peripheral neuropathy (NCI CTC AE v4.0), grade II or above congestive heart failure (NCI CTC AE v4.0), myocardial infarction in 6 month, thyroid dysfunction (> level 2 of NCI - CTC AE v4.0), etc;
9. Patients with brain、dura mater metastases or history of psychogeny;
10. Gastrointestinal bleeding in the past six months or have clear gastrointestinal bleeding tendency,such as: patients of local active ulcerative lesions, defecate occult blood + + above shall not enter into group; defecate occult blood + depend on gastroscopy;
11. Patients with severe stomach/esophageal varices and need for intervention treatment;
12. Patients with abdominal fistula, gastrointestinal perforation or abdominal abscess within 4 weeks before the first treatment;
13. Patients with glomenrular filtration rate abnormal obviously(The endogenous creatinine clearance < 60 ml/min or serum creatinine > 1.5 x ULN);
14. Positive for HIV antibody;
15. Patients who are allergic to computed tomography (CT) and magnetic resonance imaging (MRI) contrast agents at the same time, can't imaging assay;
16. Patients accepted any experimental drugs or pilot medical apparatus and instruments in the past 4 weeks of first treatment;
17. Other reasons the researchers think not suitable.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-01-27 (Estimated); Study Completion 2021-01-28 (Estimated)

PRIMARY OUTCOMES:
OS | 3 years
  Overrall survival.The time of patient from randomization to death caused by any cause.

SECONDARY OUTCOMES:
PFS | 3 years
  Progression-free survival.The time of patients from randomization to death caused by the progression of the tumor or any cause.
TTP | 1 years
  Time tumor progression.The time of patient from randomization to objective progress of the tumor.
DCR | 1 years
  Disease control rate.The proportion of patients who had a best response rating of complete response, partial response, or stable disease.
ORR | 1 years
  Objective response rate.The proportion of patients who had a best response rating of complete response and partial response.
SRR | 1 years
  Symptom remission rate. The proportion of symptoms are alleviated in all evaluative cases.

CONTACTS AND LOCATIONS:
Overall Officials: Yinying Lu, Doctor, Study Director — Liver Cancer Diagnosis & Treatment and Research Center of 302 Military Hospital of China
Locations (1):
- 302 Military Hospital of China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: When the study is finished